CLINICAL TRIAL: NCT06046183
Title: Outcomes of Small Group Process Work on Medical Students' Resilience, Grit, and Stress Over Multiple Cohorts
Brief Title: Resilience, Grit, and Stress in Medical Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Principal Investigator, Edie Sperling, Assistant Professor and Vice-Chair, Medical Anatomical Sciences, Western University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1902099-2
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Stress, Psychological
Keywords: medical students; resilience; grit; stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Control group and intervention group who self-selects
Who Masked: Care Provider
Masking Description: Interventionist is blinded to which group participants are also research participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Process Group (Experimental): Medical students enrolled in the small process group, led by psychiatrist.
  Interventions: Behavioral: Process group
- Control Group (No Intervention): Medical students from the same cohorts, not enrolled in the small process group.

INTERVENTIONS:
Behavioral: Process group — The medical student process group serves as a space for students to gain increased self-awareness through guided exploration of the psychodynamic processes.
  Arms: Process Group

SUMMARY:
The incidence of burnout and mental ill-health begins very early in medical school and continues to be high throughout training. Medical students are under high amounts of stress, which often becomes chronic, and can lead to both physical and psychological issues as a student, resident, and physician. Chronic stress and burnout in medical students are not a new phenomenon, but recent research has highlighted the worsening mental health of medical students, with as high as three-quarters of students reporting mental ill-health. It is vital that ways are found to reduce burnout and assist in improving the mental health of medical students. This quasi-experimental study is an ongoing study which is enrolling cohorts of students as they enter medical school.

DETAILED DESCRIPTION:
The investigators will assess the effects of a year-long small process group intervention, led by a psychiatrist, which aims to improve self-awareness, mindfulness, and resilience in first and second-year medical students. Students self-select into the process group, and a similar number are randomly recruited as controls from the rest of the preclinical student body. The psychiatrist is blinded to student participation in the study. Students in the process and control groups will be surveyed with the Perceived Stress Scale, the Connor-Davidson Resilience Scale, and the Grit Scale in September 2023, and again after nine months and 25 sessions, in May 2024, after the academic year. Statistical analysis will be done with R Studio. Bandura's theory of self-efficacy was used to conceptualize the study. Recruitment is done by email, as is data collection. The intervention includes guided exploration of the psychodynamic process, group dynamic theory, cognitive behavioral therapy, dialectical behavioral therapy, boundaries, and empathy.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be an enrolled student at the College of Osteopathic Medicine of the Pacific-NW
2. Participant must be in their first or second year of medical school
3. Participant must be at least 18 years of age
4. Participant must self-select into either the intervention group or control group
5. Participant must sign informed consent

Exclusion Criteria:

1. Data will be excluded if a student goes on a LOA during the course of the year
2. Data will be excluded if a student does not attend a minimum of 12 out of 25 small group sessions
3. Student does not give informed consent
4. Student withdraws consent at any time

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale-14 | 34 weeks
  Stress measured on a 0-56 scale; higher number means more stress. Each of the 14 questions is measured on a 0-4 scale of 0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often.
Connor-Davidson Resilience Scale-25 | 34 weeks
  Resilience is measured on this 25-item scale, with higher numbers meaning more resilience. The score can range between 0 and 100. Each item has anchors from 0-4.
The Grit Scale | 34 weeks
  The original 12-item grit scale was used to measure grit; each items is rated 1-5, then scores are summed and divided by 12, so the final score is between 1-5. Higher scores mean more grit.

SECONDARY OUTCOMES:
Medication or diagnosis change | 34 weeks
  Change in anti-depression, anti-anxiety, or other mental health medications or diagnoses on a binary yes/no scale.

CONTACTS AND LOCATIONS:
Overall Officials: Edie Sperling, DPT, Principal Investigator — Western University of Health Sciences
Locations (1):
- Western University of Health Science, College of Osteopathic Medicine of the Pacific - Northwest, Lebanon, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All anonymized demographic and outcome data will be shared in an open-access data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after being received and cleaned after the second timepoint in May 2024
Access Criteria: Data will be open access